CLINICAL TRIAL: NCT02860013
Title: Effectiveness and Cost-effectiveness of Telemedicine for Heart Failure: The Danish "TeleCare North" Pragmatic Randomized Trial
Brief Title: Telemedicine for Patients Suffering From Heart Failure (Danish Telecare North Trial)
Acronym: TCN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University (Other)
Responsible Party: Principal Investigator, Ole K. Hejlesen, Professor, Aalborg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: telecare nord heart failure
Record Dates: First submitted 2016-07-28; First posted 2016-08-09 (Estimated); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Heart Failure
Keywords: Telemedicine; Effectiveness; Cost-effectiveness
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telemedicine (Active Comparator): A tablet (a Samsung GALAXY TAB 2 (10.1)) that holds information on handling heart failure in general. The device can also collect and transmit relevant disease-specific data, which are indicative of their current state of health, via a Digital Blood Pressure Monitor (Model UA-767, plus BT-C) and a scale. The device can measure four vital signs, which are transferred wirelessly: blood pressure, pulse, and weight. The tablet can be activated and give a sound, when it is time for taking measurements again.
  Interventions: Device: Telemedicine
- Usual care (No Intervention): In Denmark, usual practice for treating, monitoring and caring for patients with heart failure are the responsibility of the patient's general practitioner (treatment and monitoring) and the municipalities (practical help and nursing care). Heart failure patients can make appointments with their general practitioner or practice nurse free of charge in order to get help in managing heart failure. Community based care and practical help varies. As a rule community care comes at regular intervals based on a clinically based estimate of the patients' needs, but the personnel are not necessarily certified nurses and often not fully educated in heart failure and definitely not on call

INTERVENTIONS:
Device: Telemedicine
  Arms: Telemedicine

SUMMARY:
There are two main aims in this study. The first objective is to evaluate whether a particular telehealth solution, in addition to standard treatment and care, lead to a significant decrease in the mortality and an increase in health related quality of life for patients suffering from Heart Failure that may benefit from telehealth compared with only standard treatment and care. The second objective is to examine the additional costs of the telehealth solution and assess whether this solution is a cost-effective way to care for patients with Heart Failure across patients and municipality districts.

It is hypothesized that telehealth care will increase patients quality adjusted life years compared to usual practice, since no difference in mortality and a higher health related quality of life is expected. Furthermore, it is hoped that there will be a 30% reduction in the number of admissions and readmissions to hospitals and a 30% reduction in the number of outpatient visits resulting in fewer costs for hospitals. However, it is uncertain as to whether these savings are offset by other costs such as more visits to general practitioners, community care or the implementation costs.

ELIGIBILITY:
Inclusion Criteria:

* All heart failure patients that may benefit from telehealthcare.
* Participants are qualified for inclusion if they have been diagnosed with HF according to national guidelines and are NYHA classified 2,3, and 4.
* Patients must have a permanent residence and be motivated for using telehealthcare. *Patients must have a landline or mobile phone and be able to speak Danish or they must live with a relative speaking Danish. Such that the relative must be able to help the patient in translating the information in the use of telehealthcare.

Exclusion Criteria:

* Patients without landline phone / mobile phone or GSM (Global System for Mobile Communications) coverage.
* Patients not able to understand Danish adequately to complete the questionnaires in the study or patients having a cognitive impairment.
* Comorbidity is not an exclusion criterion.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2016-08; Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

PRIMARY OUTCOMES:
Mental health related quality of life (SF-36 questionnaire mental scores) | 12 month follow-up
  Changes in mental health-related quality of life (SF-36 questionnaire mental score) at baseline to follow-up.
Incremental cost-effectiveness ratio (ICER) | 12 month follow-up
  The main outcome for cost is incremental cost-effectiveness ratio (ICER). ICER is measured as the total cost per quality adjusted life years (QALY) increased from baseline to follow-up.

SECONDARY OUTCOMES:
Changes in daily functioning (KCCQ questionnaire score) | 12 month follow-up
  Changes in daily functioning measured by KCCQ questionnaire score.
Physical health related quality of life (SF-36 questionnaire Physical scores) | 12 month follow-up
  Changes in physical health-related quality of life (SF-36 questionnaire physical score) at baseline to follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Aalborg University, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vestergaard AS, Hansen L, Sorensen SS, Jensen MB, Ehlers LH. Is telehealthcare for heart failure patients cost-effective? An economic evaluation alongside the Danish TeleCare North heart failure trial. BMJ Open. 2020 Jan 27;10(1):e031670. doi: 10.1136/bmjopen-2019-031670. PMID 31992604
- [Derived] Cichosz SL, Udsen FW, Hejlesen O. The impact of telehealth care on health-related quality of life of patients with heart failure: Results from the Danish TeleCare North heart failure trial. J Telemed Telecare. 2020 Aug-Sep;26(7-8):452-461. doi: 10.1177/1357633X19832713. Epub 2019 Apr 11. PMID 30975047
- [Derived] Cichosz SL, Ehlers LH, Hejlesen O. Health effectiveness and cost-effectiveness of telehealthcare for heart failure: study protocol for a randomized controlled trial. Trials. 2016 Dec 12;17(1):590. doi: 10.1186/s13063-016-1722-5. PMID 27955682